CLINICAL TRIAL: NCT00387244
Title: Efficacy of the Precision Spinal Cord Stimulation System as Salvage Therapy for Patients With Chronic Intractable Pain of the Trunk and or Limbs Who Have Failed Treatment With an Intraspinal Infusion Pump or Other Spinal Cord Stimulation Device
Brief Title: Efficacy of the Spinal Cord Stimulation System as Salvage Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Data Collected
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS0506
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Pain; Intractable Pain; Chronic Pain
Keywords: Pain; Back Pain; Neurostimulation
MeSH Terms: conditions — Pain; Pain, Intractable; Chronic Pain; Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Precision for Spinal Cord Stimulation (Experimental): Single arm Precision for Spinal Cord Stimulation
  Interventions: Device: Precision for Spinal Cord Stimulation

INTERVENTIONS:
Device: Precision for Spinal Cord Stimulation — Precision System aids in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, intractable back pain, and leg pain.
  Other Names: PRECISION Spinal Cord Stimulator System (Precision System)

SUMMARY:
The primary objective of this study is to evaluate the efficacy of spinal cord stimulation using the Precision implantable neurostimulation device for chronic and intractable pain of the trunk and or limbs in patients who have failed treatment with an intraspinal infusion pump or other SCS system.

DETAILED DESCRIPTION:
Chronic pain is managed by the sequential application of various strategies: medications, anesthetic injections, ablation, surgery, implantable intraspinal infusion pumps, and spinal cord stimulation. For a significant number of patients, however, these treatments are inadequate or cannot be tolerated. Those patients require another option for pain relief.

The therapy afforded by spinal cord stimulators is dependent on overlapping paresthesia with the painful areas. One of the leading reasons for explant of SCS systems (not including device failure or surgical complication) is the complaint of inadequate pain relief due to poor coverage of the painful area. Mounting evidence suggests that the clinical efficacy afforded by SCS varies with each manufacturer's technology. For instance, previously-implanted SCS patients report more complete coverage, better pain relief, and a more pleasant sensation associated with the paresthesia of the Precision system. The tight lead spacing and current fractionalization achievable with the Precision system may provide pain relief after failure with another SCS system.

This study will assess pain relief with the Precision system for patients with chronic, intractable pain who are refractory to treatment with other types of SCS systems and/or implantable intraspinal infusion pumps. Because Precision allows unique programming combinations not possible with other systems, it is expected that subjects will enjoy significant pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic and intractable neuropathic pain of the trunk and/or limbs of moderate to severe intensity and have failed treatment with an intraspinal infusion pump or other SCS device. Determination of failure of treatment will be based on subject feedback. Subjects with an active intraspinal infusion pump but with inadequate pain control will be allowed to participate;
* Be 18 years of age or older;
* Be an appropriate candidate for the surgical procedures required for this study;
* Be willing and able to comply with all study related procedures and visits;
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have failed immediate past treatment with an intraspinal infusion pump or other SCS device because of technical reasons associated with the device such as unresolved lead migration, battery depletion, etc.;
* Have any evidence of neurologic instability requiring surgery;
* Have any significant medical condition that in the opinion of the investigator may interfere with the conduct of the study or may adversely affect the subject's safety during the study;
* Have any other active implantable device with the exception of a intraspinal infusion pump for pain medications;
* Are pregnant or lactating or planning to become pregnant in the next year;
* Have participated in any investigational drug or device trial in the last 4 weeks or plan to participate in any other investigational drug or device trial while on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (1):
- Spectrum Care, Napa, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Precision for Spinal Cord Stimulation
Started | 7
End of Trial | 0
Completed | 0
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Precision for Spinal Cord Stimulation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With a Significant Reduction in Pain During the Temporary Trial
Time Frame: Baseline and at End of trial (approximately 5 days)
Population: The study was terminated and efforts were made to locate data. No study data are available.
Arm/Group | Precision for Spinal Cord Stimulation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through completion of data collection (26 weeks post-activation or withdrawal).
Description: Insufficient data
Arm/Group | Precision for Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Insufficient data collected to report results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes